CLINICAL TRIAL: NCT05911061
Title: A Multicenter, Randomized, Double-Blind, Controlled, Phase Ⅲ Clinical Trial of Recombinant COVID-19 Trivalent (XBB+BA.5+Delta) Protein Vaccine (Sf9 Cell) in Booster Vaccination to Evaluate Efficacy, Safety and Immunogenicity in Population Aged 18 Years Old and Above
Brief Title: A Phase Ⅲ Clinical Trial of Recombinant COVID-19 Trivalent (XBB+BA.5+Delta) Protein Vaccine (Sf9 Cell) in Booster Vaccination
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: WestVac Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WSKCT015
Record Dates: First submitted 2023-06-19; First posted 2023-06-20 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental group 1 (Experimental): high dose
  Interventions: Biological: High dose of Recombinant COVID-19 Trivalent (XBB+BA.5+Delta) Protein Vaccine (Sf9 Cell)
- Experimental group 2 (Experimental): low dose
  Interventions: Biological: Low dose of Recombinant COVID-19 Trivalent (XBB+BA.5+Delta) Protein Vaccine (Sf9 Cell)
- Control group (Active Comparator): Control group
  Interventions: Biological: control group
- Placebo control group (Placebo Comparator): Placebo control group
  Interventions: Biological: Placebo group

INTERVENTIONS:
Biological: High dose of Recombinant COVID-19 Trivalent (XBB+BA.5+Delta) Protein Vaccine (Sf9 Cell) — boost with high dose of Recombinant COVID-19 Trivalent (XBB+BA.5+Delta) Protein Vaccine (Sf9 Cell)
  Arms: Experimental group 1
Biological: Low dose of Recombinant COVID-19 Trivalent (XBB+BA.5+Delta) Protein Vaccine (Sf9 Cell) — boost with low dose of Recombinant COVID-19 Trivalent (XBB+BA.5+Delta) Protein Vaccine (Sf9 Cell)
  Arms: Experimental group 2
Biological: control group — boost with Recombinant Variant COVID-19 Vaccine(sf9 cell)
  Arms: Control group
Biological: Placebo group — saline
  Arms: Placebo control group

SUMMARY:
A Phase Ⅲ Clinical Trial of Recombinant COVID-19 Trivalent (XBB+BA.5+Delta) Protein Vaccine (Sf9 Cell) in Booster Vaccination to Evaluate Efficacy, Safety and Immunogenicity

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-Blind, Controlled, Phase Ⅲ Clinical Trial of Recombinant COVID-19 Trivalent (XBB+BA.5+Delta) Protein Vaccine (Sf9 Cell) in Booster Vaccination to Evaluate Efficacy, Safety and Immunogenicity in Healthy Population Aged 18 Years Old and Above

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18 years and above, including those with underlying diseases and immunocompromised subjects.
2. Basic or booster immunization with COVID-19 vaccine ≥6 months.
3. ≥3 months of SARS-CoV-2 infection history, or never infected.
4. Have the ability to understand research procedures, with informed consent, voluntarily sign informed consent, and be able to comply with the requirements of clinical research protocols.

Exclusion Criteria:

1. Axillary temperature ≥37.3℃.
2. SARS-CoV-2 antigen or nucleic acid screening positive within the last 48 hours.
3. Anti-SARS-CoV-2 IgM antibody was positive during the screening period.
4. It is in the advanced stage of malignant tumor and the disease control is unstable.
5. Female pregnancy (pregnancy test results are positive), lactation period.
6. Have serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, heart failure, severe hypertension, and can not be controlled by drugs.
7. Have other serious chronic conditions such as uncontrolled asthma, diabetes, chronic obstructive pulmonary disease, pulmonary embolism, chronic kidney disease requiring dialysis, cirrhosis of the liver, convulsions, epilepsy and other neurological/psychiatric conditions.
8. Have been diagnosed with congenital or acquired immunodeficiency, HIV infection.
9. People who are allergic to any component of the investigational vaccine have a history of more severe allergies or allergic reactions to the vaccine in the past.
10. Congenital or acquired angioedema/neuroedema.
11. Asplenia or functional asplenia.
12. Thrombocytopenia or other clotting disorders (which may cause intramuscular injection contraindications).
13. Received another investigational drug within 1 month prior to receiving the investigational vaccine.
14. Received subunit or inactivated vaccine within 14 days prior to receiving the investigational vaccine, or received live attenuated vaccine within 1 month.
15. Fertile female subjects did not use effective contraception within 1 month prior to enrollment.
16. Fertile female and male subjects have pregnancy plans and sperm/egg donation plans from the screening period to 3 months after immunization.
17. Abnormal laboratory test results during the screening period, which were judged by the researcher to be unsuitable for the study vaccine.
18. Medical, psychological, social, or other conditions that, in the investigator's judgment, are inconsistent with the protocol or affect the subject's signing of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4950 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy against COVID-19 | 14 days after vaccination
  Efficacy against the first occurrence of a virologically confirmed (PCR-positive) case of symptomatic COVID-19, regardless of severity, 14 days after booster vaccination.
AE and AR | 0-7 days after vaccination
  Incidence of adverse events (AE) and adverse reactions (AR) 0-7 days after booster vaccination.

SECONDARY OUTCOMES:
Secondary Efficacy against COVID-19 | >7 days after booster vaccination
  Efficacy against the first occurrence of a virologically confirmed (PCR-positive) case of symptomatic COVID-19 > 7 days after booster vaccination in subjects, regardless of severity.
Secondary Efficacy against COVID-19 | > 7 days and > 14 days after booster vaccination
  Efficacy against first occurrence of virologically confirmed (PCR-positive) cases of moderate/severe COVID-19 caused by SARS-CoV-2 infection, cases of hospitalization due to COVID-19, and cases of death due to COVID-19, > 7 days and > 14 days after booster vaccination
Secondary Safety | 0-30 days after booster vaccination
  Incidence of adverse events (AE) and adverse reactions (AR) 0-30 days after booster vaccination.
Secondary Safety | within 12 months after booster vaccination
  Incidence of serious adverse events (SAE) and adverse events of special interest (AESI) within 12 months after booster vaccination.
Secondary Immunogenicity indicator 1 | day 14, day 30 and 3 months after booster vaccination
  The geometric mean titer (GMT), seroconversion rate and geometric mean fold increase (GMI) of neutralizing antibodies against SARS-CoV-2 variants (based on the current variants at same time) on day 14, day 30 and 3 months after booster vaccination.
Secondary Immunogenicity indicator 2 | day 14, day 30 and 3 months after booster vaccination
  Geometric mean titer (GMT), seroconversion rate and geometric mean fold increase (GMI) of anti-SARS-CoV-2 specific binding antibodies were measured on day 14, day 30 and 3 months after booster vaccination.